CLINICAL TRIAL: NCT05288478
Title: Phase II Dose-ranging Study of Dentoxol® Mouthrinse for Managing Oral Symptoms in Epidermolysis Bullosa.
Brief Title: Dose-ranging Study of Dentoxol® Mouthrinse for Managing Oral Symptoms in People With Epidermolysis Bullosa.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Chile (Other)
Collaborators: Fundación DEBRA Chile, Niños Piel de Cristal (Other)
Responsible Party: Principal Investigator, Susanne Kramer, Associate Professor, University of Chile
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: PRI-ODO 2021/16
Record Dates: First submitted 2021-11-24; First posted 2022-03-21 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Epidermolysis Bullosa; Oral Ulcer
Keywords: Epidermolysis Bullosa; Oral ulcer; Oral blisters; Dentoxol mouthrinse
MeSH Terms: conditions — Epidermolysis Bullosa; Oral Ulcer

STUDY DESIGN:
Intervention Model Description: 100 subjects with EB will be recruited, divided into groups according to their mayor type of EB and subtype, they will use Dentoxol® mouthrinse twice a day or 5 times each day.
  Subjects will have a dose regimen assigned randomly, group A: first 6 weeks 5 times a day, following 6 weeks twice a day, and group B: first 6 weeks 2 times a day following 6 weeks 5 times a day, both with a 4 week washout period in between.
  On week 0, 1, 3 and 6 of each regime patients living in the metropolitan area will be examined by the Oral Medicine specialist.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group A (Active Comparator): First 6 weeks they will use the mouthrinse 5 times a day, following 4 week washout period.
  Interventions: Combination Product: Dentoxol mouthrinse dosages
- Group A, second period (Active Comparator): After the washout period, the next 6 weeks the will use the mouthrinse twice a day.
  On week 0, 1, 3 and 6 of each regime patients living in the metropolitan area will be examined by the Oral Medicine specialist.
  Interventions: Combination Product: Dentoxol mouthrinse dosages
- Group B (Active Comparator): First 6 weeks they will use the mouthrinse twice a day, following 4 week washout period
  Interventions: Combination Product: Dentoxol mouthrinse dosages
- Group B, second period (Active Comparator): After the washout period, the next 6 weeks they will use the mouthrinse 5 times a day.
  On week 0, 1, 3 and 6 of each regime patients living in the metropolitan area will be examined by the Oral Medicine specialist.
  Interventions: Combination Product: Dentoxol mouthrinse dosages

INTERVENTIONS:
Combination Product: Dentoxol mouthrinse dosages — Subjects will have a dose regimen assigned randomly, group A: first 6 weeks 5 times a day, following 6 weeks twice a day, and group B: first 6 weeks 2 times a day following 6 weeks 5 times a day, both with a 4 week washout period in between.

SUMMARY:
Inherited Epidermolysis Bullosa (EB) is a disorder that causes skin fragility and blistering in skin and mucous membranes, including the mouth. Recurrent oral blisters and ulcer result in oral pain and discomfort.

Dentoxol® is a mouthrinse that has anti-inflammatory, antimicrobial and analgesic effects. It has significant potential to reduce EB related oral symptoms.

This study includes people living with Inherited Epidermolysis Bullosa aged 6 and above; and is aimed at determining the efficacy of two different dose regimens of Dentoxol mouthrinse in reducing oral symptoms.

DETAILED DESCRIPTION:
Inherited Epidermolysis Bullosa (EB) is a group of genetic disorders with skin fragility and blistering. In addition to the skin, it can affect the mucous membranes, causing oral symptoms including oral pain and discomfort due to recurrent oral blisters, ulcers and erosions. Dentoxol® is a proprietary mouthrinse that has anti-inflammatory, antimicrobial and analgesic effects. This three-pronged strategy therefore has significant potential to reduce EB related oral symptoms.

Preliminary reports of Dentoxol® mouthrinse have suggested that it is safe and effective in reducing the EB related oral symptoms.Therefore, a well-controlled Phase II study is now warranted.

This study will include people living with Inherited Epidermolysis Bullosa aged 6 and over, and seeks to determinate the efficacy of two different dose regimens of Dentoxol mouthrinse in reducing the symptoms mentioned above.

Methods: 100 subjects with EB will be recruited and will be given Dentoxol® mouthrinse for two periods of 6 weeks using different dose regimes.

Subjects will have a dose regimen assigned randomly, group A: first 6 weeks will be asked to rinse 5 times a day, followed by a 4 weeks washout period and the second 6 weeks period: twice a day. Group B: first 6 weeks 2 times a day, second 6 weeks period: 5 times a day, both with a 4 week washout period in between.

On week 0, 1, 3 and 6 of each regime patients living in the metropolitan area will be examined by the Oral Medicine specialist.

ELIGIBILITY:
Inclusion Criteria:

* People living with Inherited Epidermolysis Bullosa, including all types and subtypes, registered at Debra Foundation at the country of the study.

Exclusion Criteria:

* Unable to give written informed consent / assent.
* Have used a mouth rinse aimed at managing oral ulcers in the last 4 weeks.
* Known allergy/intolerance to any component of the study rinse.
* Planning to use any of the following contraindicated medications during the study period (pain medications are allowed)
* Any agent marketed for oral mucositis
* Steroids
* Antibiotics (eg, tetracyclines) (Note: topical antifungals are allowed)
* Povidone iodine
* Sucralfate and other coating agents such as Gelclair, MuGard, etc.
* Caphosol
* Chlorhexidine Gluconate (Oralgene, Perioaid, Peridex, Periogard)
* Diphenhydramine (Benadryl)
* Laser therapy for oral mucositis
* Any other anti-inflammatory agent
* Any other investigative agent
* *Note: "Miracle / Magic" rinse preparations containing viscous lidocaine are allowed, however, diphenhydramine and other excluded agents should not be added.
* Age below 6 years
* Pregnant or nursing
* Unable to rinse the mouth due to limited oral functioning.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-04-06 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Change in oral symptoms associated to oral bullae, erosions and ulcerations in adults and children over the age of 6 living with Epidermolysis Bullosa with two different dose regimes of Dentoxol® mouthrinse and compare both effects. | 16 weeks
  Epidermolysis Bullosa Oral Health Questionnaire (EBOHQ)

SECONDARY OUTCOMES:
Change in the duration of the lesions with two different dose regimes of Dentoxol® mouthrinse and compare both effects. | 16 weeks
  Epidermolysis Bullosa Oral Health Questionnaire (EBOHQ) (Validated Questionnaire)
Change in the frequency of the lesions with two different dose regimes of Dentoxol® mouthrinse and compare both effects. | 16 weeks
  Epidermolysis Bullosa Oral Health Questionnaire (EBOHQ) (Validated Questionnaire)
Change in the recurrence of the lesions with two different dose regimes of Dentoxol® mouthrinse and compare both effects. | 16 weeks
  Epidermolysis Bullosa Oral Health Questionnaire (EBOHQ) (Validated Questionnaire)
Change in the size of the lesions with two different dose regimes of Dentoxol® mouthrinse and compare both effects. | 16 weeks
  Epidermolysis Bullosa Oral Health Questionnaire (EBOHQ) (Validated Questionnaire)
Change in the number of the lesions with two different dose regimes of Dentoxol® mouthrinse and compare both effects. | 16 weeks
  Epidermolysis Bullosa Oral Health Questionnaire (EBOHQ) (Validated Questionnaire)
Change in the distribution of the lesions with two different dose regimes of Dentoxol® mouthrinse and compare both effects. | 16 weeks
  Epidermolysis Bullosa Oral Health Questionnaire (EBOHQ) (Validated Questionnaire)
Change in oral pain with two different dose regimes of Dentoxol® mouthrinse and compare both effects. | 16 weeks
  Epidermolysis Bullosa Oral Health Questionnaire (EBOHQ) (Validated Questionnaire)
Improve the oral health related quality of life and oral functioning with two different dose regimes of Dentoxol® mouthrinse and compare both effects. | 16 weeks
  Epidermolysis Bullosa Oral Health Questionnaire (EBOHQ) (Validated Questionnaire)
Patients compliance with treatment. | 16 weeks
  Daily record of mouthrinse use.
Patients acceptance of mouthrinse use | 16 weeks
  Mouthrinse Acceptance Form (Validated Questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Kramer, MsC, Principal Investigator — University of Chile
Locations (1):
- Facultad de Odontología, Universidad de Chile, Santiago, Santiago Metropolitan, Chile

REFERENCES:
- [Background] Has C, Bauer JW, Bodemer C, Bolling MC, Bruckner-Tuderman L, Diem A, Fine JD, Heagerty A, Hovnanian A, Marinkovich MP, Martinez AE, McGrath JA, Moss C, Murrell DF, Palisson F, Schwieger-Briel A, Sprecher E, Tamai K, Uitto J, Woodley DT, Zambruno G, Mellerio JE. Consensus reclassification of inherited epidermolysis bullosa and other disorders with skin fragility. Br J Dermatol. 2020 Oct;183(4):614-627. doi: 10.1111/bjd.18921. Epub 2020 Mar 11. PMID 32017015
- [Background] Uitto J. Toward treatment and cure of epidermolysis bullosa. Proc Natl Acad Sci U S A. 2019 Dec 26;116(52):26147-26149. doi: 10.1073/pnas.1919347117. Epub 2019 Dec 11. No abstract available. PMID 31826952
- [Background] Has C, Liu L, Bolling MC, Charlesworth AV, El Hachem M, Escamez MJ, Fuentes I, Buchel S, Hiremagalore R, Pohla-Gubo G, van den Akker PC, Wertheim-Tysarowska K, Zambruno G. Clinical practice guidelines for laboratory diagnosis of epidermolysis bullosa. Br J Dermatol. 2020 Mar;182(3):574-592. doi: 10.1111/bjd.18128. Epub 2019 Aug 9. PMID 31090061
- [Background] Korolenkova MV. [Dental treatment in children with dystrophic form of epidermolysis bullosa]. Stomatologiia (Mosk). 2015;94(2):34-36. doi: 10.17116/stomat201594234-36. Russian. PMID 26145475
- [Background] Puliyel D, Chiu CH, Habibian M. Restorative and periodontal challenges in adults with dystrophic epidermolysis bullosa. J Calif Dent Assoc. 2014 May;42(5):313-8. PMID 25087349
- [Background] Mello BZ, Neto NL, Kobayashi TY, Mello MB, Ambrosio EC, Yaedu RY, Machado MA, Oliveira TM. General anesthesia for dental care management of a patient with epidermolysis bullosa: 24-month follow-up. Spec Care Dentist. 2016 Jul;36(4):237-40. doi: 10.1111/scd.12170. Epub 2016 Mar 2. PMID 26936632
- [Background] Pekiner FN, Yucelten D, Ozbayrak S, Sezen EC. Oral-clinical findings and management of epidermolysis bullosa. J Clin Pediatr Dent. 2005 Fall;30(1):59-65. doi: 10.17796/jcpd.30.1.y503845545kn78x7. PMID 16302602
- [Background] Oliveira TM, Sakai VT, Candido LA, Silva SM, Machado MA. Clinical management for epidermolysis bullosa dystrophica. J Appl Oral Sci. 2008 Jan-Feb;16(1):81-5. doi: 10.1590/s1678-77572008000100016. PMID 19089295
- [Background] Kummer TR, Nagano HC, Tavares SS, Santos BZ, Miranda C. Oral manifestations and challenges in dental treatment of epidermolysis bullosa dystrophica. J Dent Child (Chic). 2013 May-Aug;80(2):97-100. PMID 24011299
- [Background] Marini I, Vecchiet F. Sucralfate: a help during oral management in patients with epidermolysis bullosa. J Periodontol. 2001 May;72(5):691-5. doi: 10.1902/jop.2001.72.5.691. PMID 11394407
- [Background] Fortuna G, Lozada-Nur F, Pollio A, Aria M, Cepeda-Valdes R, Marinkovich MP, Bruckner AL, Salas-Alanis JC. Patterns of oral mucosa lesions in patients with epidermolysis bullosa: comparison and agreement between oral medicine and dermatology. J Oral Pathol Med. 2013 Nov;42(10):733-40. doi: 10.1111/jop.12094. Epub 2013 Jun 15. PMID 23772832
- [Background] Fortuna G, Aria M, Cepeda-Valdes R, Pollio A, Moreno-Trevino MG, Salas-Alanis JC. Clinical features of gingival lesions in patients with dystrophic epidermolysis bullosa: a cross-sectional study. Aust Dent J. 2015 Mar;60(1):18-23. doi: 10.1111/adj.12264. PMID 25721275
- [Background] Brun J, Chiaverini C, Devos C, Leclerc-Mercier S, Mazereeuw J, Bourrat E, Maruani A, Mallet S, Abasq C, Phan A, Vabres P, Martin L, Bodemer C, Lagrange S, Lacour JP; Research Group of the French Society of Pediatric Dermatology. Pain and quality of life evaluation in patients with localized epidermolysis bullosa simplex. Orphanet J Rare Dis. 2017 Jun 28;12(1):119. doi: 10.1186/s13023-017-0666-5. PMID 28659151
- [Background] Stellingsma C, Dijkstra PU, Dijkstra J, Duipmans JC, Jonkman MF, Dekker R. Restrictions in oral functions caused by oral manifestations of epidermolysis bullosa. Eur J Dermatol. 2011 May-Jun;21(3):405-9. doi: 10.1684/ejd.2011.1356. PMID 21609900
- [Background] Wright JT. Comprehensive dental care and general anesthetic management of hereditary epidermolysis bullosa. A review of fourteen cases. Oral Surg Oral Med Oral Pathol. 1990 Nov;70(5):573-8. doi: 10.1016/0030-4220(90)90401-d. PMID 2146579
- [Background] Cheng KK. Children's acceptance and tolerance of chlorhexidine and benzydamine oral rinses in the treatment of chemotherapy-induced oropharyngeal mucositis. Eur J Oncol Nurs. 2004 Dec;8(4):341-9. doi: 10.1016/j.ejon.2004.04.002. PMID 15550364
- [Background] Sindici E, Astesano S, Fazio L, Dragonetti A, Pugliese M, Scully C, Carossa S, Broccoletti R, Arduino PG. Treatment of Oral Lesions in Dystrophic Epidermolysis Bullosa: A Case Series of Cord Blood Platelet Gel and Low-level Laser Therapy. Acta Derm Venereol. 2017 Mar 10;97(3):383-384. doi: 10.2340/00015555-2512. No abstract available. PMID 27535037
- [Background] Kramer S, Lucas J, Gamboa F, Penarrocha Diago M, Penarrocha Oltra D, Guzman-Letelier M, Paul S, Molina G, Sepulveda L, Araya I, Soto R, Arriagada C, Lucky AW, Mellerio JE, Cornwall R, Alsayer F, Schilke R, Antal MA, Castrillon F, Paredes C, Serrano MC, Clark V. Clinical practice guidelines: Oral health care for children and adults living with epidermolysis bullosa. Spec Care Dentist. 2020 Nov;40 Suppl 1(Suppl 1):3-81. doi: 10.1111/scd.12511. PMID 33202040
- [Background] Lalla RV, Sole S, Becerra S, Carvajal C, Bettoli P, Letelier H, Santini A, Vargas L, Cifuentes A, Larsen F, Jara N, Oyarzun J, Feinn R, Bustamante E, Martinez B, Rosenberg D, Galvan T. Efficacy and safety of Dentoxol(R) in the prevention of radiation-induced oral mucositis in head and neck cancer patients (ESDOM): a randomized, multicenter, double-blind, placebo-controlled, phase II trial. Support Care Cancer. 2020 Dec;28(12):5871-5879. doi: 10.1007/s00520-020-05358-4. Epub 2020 Apr 8. PMID 32266567
- [Derived] Rojas P, Kramer S, Veliz S, Seguel M, Alsayer F, Sepulveda L. Dentoxol Mouthwash for People With Epidermolysis Bullosa: A Qualitative Study of Self-Perceived Symptoms and Quality of Life. Spec Care Dentist. 2025 Mar-Apr;45(2):e70036. doi: 10.1111/scd.70036. PMID 40268883